CLINICAL TRIAL: NCT01110421
Title: A Prospective, Randomized, Double-Blind, Multicenter Study to Establish the Safety and Tolerability of Doripenem Compared With Cefepime in Hospitalized Children With Bacterial Pneumonia
Brief Title: A Safety and Tolerability Study of Doripenem Compared With Cefepime in Hospitalized Children With Bacterial Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial terminated early per business decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016975; DORIPED3003 (Other: Janssen Research & Development, LLC); 2009-016069-27 (EudraCT Number)
Record Dates: First submitted 2010-04-15; First posted 2010-04-26 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Pneumonia, Bacterial; Community-Acquired Infections; Nosocomial Infection; Pneumonia, Ventilator-Associated
Keywords: Doripenem; Child, Hospitalized; Cefepime; Infusions, Intravenous; Severe community acquired pneumonia; Nosocomial pneumonia; Ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Infections; Cross Infection; Pneumonia, Ventilator-Associated; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia | interventions — Cefepime; Doripenem; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doripenem (Experimental): Doripenem 20 mg/kg per dose (up to 500 mg/dose) will be administered every 8 hours as 60-minutes IV (at least 3 days of IV doripenem only or IV doripenem followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
  Interventions: Drug: Cefepime placebo; Drug: Doripenem; Drug: Amoxicillin/clavulanate potassium
- Cefepime (Experimental): Cefepime 50 mg/kg per dose (up to 2 g/dose) will be administered every 8 hours as 30-minutes IV (at least 3 days of IV cefepime only or IV cefipime followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
  Interventions: Drug: Cefepime; Drug: Doripenem placebo; Drug: Amoxicillin/clavulanate potassium

INTERVENTIONS:
Drug: Cefepime placebo — Form=solution for infusion, Route=intravenous use, administered once every 8 hours infused over 30 minutes immediately before each iv infusion of doripenem for up to 14 days
  Arms: Doripenem
Drug: Cefepime — Type=once every 8 hours, Unit=mg, Number=50 mg/kg up to 2g/dose, Form=solution for infusion, Route=intravenous use. At least 3 days of iv cefepime administered every 8 hours infused over 30 minutes immediately before each iv infusion of doripenem placebo for up to 14 days
  Arms: Cefepime
Drug: Doripenem — Type=once every 8 hours infused over 60 minutes, Unit=mg, Number=20mg/kg up to 500mg/dose, Form=solution for infusion, Route=intravenous use. At least 3 days of iv doripenem administered every 8 hours immediately after each iv infusion of cefepime placebo for up to 14 days
  Arms: Doripenem
Drug: Doripenem placebo — Form=solution for infusion, Route=intravenous use, administered once every 8 hours infused over 60 minutes immediately following each iv infusion of cefepime for up to 14 days
  Arms: Cefepime
Drug: Amoxicillin/clavulanate potassium — Form=suspension or tablets, Route=oral (by mouth), may be administered at the discretion of the investigator once every 12 hours for up to 14 days following IV therapy with doripenem or cefepime.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of doripenem compared to cefepime in children hospitalized with pneumonia.

DETAILED DESCRIPTION:
This is a randomized (study assigned by chance), double-blind (neither physician nor patient knows the name of the assigned study drugs), double-dummy (all patients will be given both a placebo [salt solution] and study drug in alternating periods of time during the study), active comparator-controlled (compare the 'test' treatment to standard-of-care therapy), multinational, multicenter study to establish the safety and tolerability of doripenem (an antibiotic) compared with cefepime (an antibiotic) administered by intravenous (iv) infusion (slow injection of drug solution into the vein over a period of time) in children ages 3 months to less than 18 years hospitalized with pneumonia (includes nosocomial pneumonia [NP], severe community-acquired pneumonia (CAP), and ventilator-assisted pneumonia [VAP]). The study includes 3 periods: a pretreatment (screening) period that will occur within 2 days prior to randomization (assignment of study drug); a treatment period of 10 to 14 days where patients will receive study drug treatment, and a posttreatment period consisting of 2 study visits. The maximum duration of study drug therapy is 14 days. The total duration of the study is approximately 7 to 8 weeks for each patient. The primary outcome measure in the study is safety and tolerability. Safety and tolerability will be evaluated by examining the incidence, severity, and type of adverse events, changes in clinical laboratory tests, vital signs measurements, and findings from physical examinations observed during treatment and at each posttreatment visit. An independent monitoring committee (IDMC) will be established for this study to ensure that the safety of the patients is not compromised. The IDMC will consist of individuals who are not associated with the conduct of the study, and will include but will not be limited to individuals with expertise relevant to the care of pediatric patients, and including at least one infectious disease physician and at least one statistician. Patients will receive IV Doripenem (20 mg/kg up to a maximum of 500 mg/dose) and cefepime placebo OR cefepime (50 mg/kg up to a maximum of 2 grams/dose and doripenem placebo once every 8 hours for up to 14 days. After receiving a minimum of 3 days of IV study drug therapy, patients may be switched to the oral antibiotic (amoxicillin/clavulanate potassium suspension or tablets) or an approved alternative oral agent to complete a total 10-14 days course of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Require parenteral antibacterial therapy for the treatment of pneumonia
* Have new or progressive radiographic infiltrate(s) (alveolar, lobar, or consolidation) consistent with a bacterial pneumonia that is not related to cardiac or other disease processes
* Must, based on the judgment of the investigator, require hospitalization initially and antibacterial therapy for 10 to 14 days for the treatment of the current pneumonia. (Note that the patient must require at least 3 days of IV antibiotic therapy initially)
* Have a diagnosis of nosocomial pneumonia , severe community-acquired pneumonia, or ventilator-associated pneumonia, defined by the disease-specific criteria as stated in the study protocol
* Have a clinical presentation compatible with bacterial pneumonia( with fever or hypothermia AND leukocytosis OR leucopenia AND at least 2 of the following clinical signs or symptoms in non-intubated patients: cough, new onset of lower respiratory tract secretions (including change in character of secretions or increase in the quantity of secretions or suctioning requirements), auscultatory findings of pneumonia or consolidation (rales, rhonchi bronchial breath sounds, decreased breath sounds, wheezing, and egophony), dyspnea, increased work of breathing expressed as retractions, nasal flaring, or grunting, hypoxemia or oxygen saturation less than 90% on room air, and tachypnea

Exclusion Criteria:

* Received more than 24 hours of systemic antibacterial therapy in the 48 hours before the start of the infusion of the first dose of study drug for the current episode of pneumonia
* Known presence at randomization of pulmonary infection caused only by bacteria that is resistant to cefepime or doripenem (including methicillin resistant Staphylococcus aureus) or presence at baseline of pulmonary infection with Stenotrophomonas species, or Burkholderia cepacia
* Has any of the following conditions at baseline that may interfere with the diagnosis or response to therapy: chest trauma with severe lung contusion, acute respiratory distress syndrome, empyema, flail chest (severe injury to the chest), history of active lung cancer, chronic bronchitis with an exacerbation within the last 30 days, bronchiectasis (an obstructive lung disease), lung abscess(s), anatomical bronchial obstruction, active pulmonary tuberculosis with treatment, suspected pulmonary tuberculosis, suspected or documented atypical viral pneumonia without bacterial superinfection, suspected or documented pertussis, chemical pneumonitis (eg, aspiration of gastric contents, inhalation injury), or cystic fibrosis
* The patient has any of the following clinically significant laboratory abnormalities: hematocrit of less than 20%
* absolute neutrophil count (ANC) <500 cells/microL, platelet count <40,000 cells/microL, serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >5x the age specific upper limit of normal, acute or chronic renal insufficiency with a baseline creatinine clearance of <60 mL/minute or requires dialysis therapy for any reason, or are profoundly immunodeficient and require prophylactic antimicrobial therapy for Pneumocystis jirovicei, Toxoplasma gondii, or herpes viruses, and/or chronic or intermittent immunoglobin replacement therapy.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (25):
- United States (4):
  - Little Rock, Arkansas
  - Cleveland, Ohio
  - Toledo, Ohio
  - Pittsburgh, Pennsylvania
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Loma Hermosa
  - Santa Fe
- Brazil (3):
  - Belo Horizonte
  - Porto Alegre
  - São Paulo
- Colombia (3):
  - Bogotá
  - Cali
  - Medellín
- Riga, Latvia
- Lithuania (3):
  - Kaunas
  - Tauragė
  - Vilnius
- Mexico (3):
  - Guadajalara
  - México
  - Monterrey
- Zona, Panama
- Poland (2):
  - Lublin
  - Szczecin
- Kharkiv, Ukraine

RESULTS

PARTICIPANT FLOW:
Groups:
- Doripenem: Doripenem 20 mg/kg per dose (up to 500 mg/dose) was administered every 8 hours as 60-minutes IV (at least 3 days of IV doripenem only or IV doripenem followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
- Cefepime: Cefepime 50 mg/kg per dose (up to 2 g/dose) was administered every 8 hours as 30-minutes IV (at least 3 days of IV cefepime only or IV cefepime followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
Period: Overall Study
Arm/Group | Doripenem | Cefepime
Started | 5 | 2
Completed | 5 (Includes 1 participant who discontinued study drug due to an adverse event of empyema on Days 9-13.) | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doripenem | Cefepime | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.2 (2.49) | 4.5 (0.71) | 5 (2.08)
Age, Customized [Number; unit: participants]
  3 months to <2 years | 0 | 0 | 0
  2 to <6 years | 3 | 2 | 5
  6 to <12 years | 2 | 0 | 2
  12 to <18 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Clinical Cure Rate at Test Of Cure (TOC) Visit
Description: The participants were classified as cure if they had resolution or clinical improvement of signs and symptoms of pneumonia, favorable response at End of treatment for IV study (EIV) visit; had no fever; improvement or no progression of radiographic findings of pneumonia on chest X ray; improvement in oxygenation or discontinued mechanical ventilation in intubated participants; and not received nonstudy systemic antibacterial therapy for pneumonia.
Time Frame: TOC (7 to 14 days after the last dose of study medication therapy)
Population: Clinical Intent-To-Treat (CITT): All randomized participants who met the minimal disease definition of pneumonia regardless if a baseline pathogen was isolated from the baseline lower respiratory tract culture, pleural fluid or blood culture.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 5 | 2
Participants | 3 | 2

2. Secondary Outcome: The Number of Participants With Clinical Improvement Rate at End of IV (EIV) Visit
Description: Participants were considered as clinical improved if they had no fever, clinical improvement in signs and symptoms of pneumonia from baseline, decrease in WBC, improvement or lack of progression of radiographic findings in comparison with the screening chest X-ray, and not received any nonstudy systemic antibacterial therapy for the treatment of pneumonia after IV study drug therapy had begun.
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy)
Population: Clinical intent-to-treat: All randomized participants who met the minimal disease definition of pneumonia regardless if a baseline pathogen was isolated from the baseline lower respiratory tract culture, pleural fluid or blood culture.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 5 | 2
Participants | 4 | 2

3. Secondary Outcome: The Number of Participants With Clinical Cure Rate at Late Follow-Up (LFU) Visit
Description: The participants were classified as clinical cure if all pretreatment signs and symptoms showed no evidence of resurgence after administration of the last dose of study medication and no nonstudy systemic antibacterial therapy was given for the treatment of pneumonia.
Time Frame: LFU (28 to 42 days after the last dose of study medication therapy)
Population: Clinical Intent-to-Treat (CITT): All randomized participants who met the minimal disease definition of pneumonia regardless if a baseline pathogen was isolated from the baseline lower respiratory tract (LRT) culture, pleural fluid or blood culture.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 5 | 2
Participants | 3 | 2

4. Secondary Outcome: The Number of Participants With Favorable Per-participant Microbiological Response Rate
Description: Favorable per-participant microbiological response rate was evaluated at the at End of IV (EIV) visit, Test Of Cure (TOC) visit, and Late Follow-Up (LFU) visit. The favorable per-participant microbiological response was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment).
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy), TOC (7 to 14 days after the last dose of study medication therapy), and LFU (28 to 42 days after the last dose of study medication therapy)
Population: Microbiological intent-to-treat - Participants of CITT with at least one baseline pneumonia pathogen from pleural fluid, LRT, or blood culture susceptible to doripenem and cefepime. 3 and 2 participants from doripenem and cefepime, respectively had no susceptible pneumonia pathogens at baseline and were excluded from this set.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 2 | 0
Participants
  TOC visit | 2 |
  EIV visit | 2 |
  LFU visit | 2 |

5. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at End of IV (EIV) Visit
Description: A total of 3 pathogens were isolated at baseline from lower respiratory tract (LRT) culture in 2 participants in the doripenem treatment group and were susceptible to the study drug received: 2 pathogens (Staphylococcus aureus Klebsiella pneumoniae) were isolated at baseline from 1 participant and a 3rd pathogen (Streptococcus pneumoniae) was isolated at baseline from the other participant (see listed in the table below; the number in parenthesis next to each pathogen represent the number of participants with the pathogen isolated at baseline in the doripenem treatment group). The favorable per-participant microbiological response was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment). NOTE: No participants in the cefepime treatment group met criteria for inclusion in the Microbiological intent-to-treat analysis.
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 2 | 0
Participants
  Staphylococcus aureus (1) | 1 |
  Streptococcus pneumoniae (1) | 1 |
  Klebsiella pneumoniae (1) | 1 |

6. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at Test Of Cure (TOC) Visit
Description: as for outcome 5
Time Frame: TOC (7 to 14 days after the last dose of study medication therapy)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 2 | 0
Participants
  Staphylococcus aureus (1) | 1 |
  Streptococcus pneumoniae (1) | 1 |
  Klebsiella pneumoniae (1) | 1 |

7. Secondary Outcome: Number of Participants With Sustained Favorable Per-pathogen Microbiological Outcome Rate at Late Follow-Up (LFU) Visit
Description: as for outcome 5
Time Frame: LFU (28 to 42 days after the last dose of study medication therapy)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 2 | 0
Participants
  Staphylococcus aureus (1) | 1 |
  Streptococcus pneumoniae (1) | 1 |
  Klebsiella pneumoniae (1) | 1 |

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks
Arm/Group | Doripenem | Cefepime
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/2
Other Adverse Events (participants affected / at risk) | 3/5 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=5) | Cefepime (N=2)
Empyema (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=5) | Cefepime (N=2)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Stab Wound (Injury, poisoning and procedural complications) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to business reasons and not related to safety concerns or issues. As such, the limited enrollment precludes a meaningful conclusion about the efficacy and safety of doripenem compared with cefepime.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days